CLINICAL TRIAL: NCT04948125
Title: Camrelizumab Combined With Apatinib for Advanced Gastric or Esophagogastric Adenocarcinoma Progressed After Immune Checkpoint Inhibitors:a Single-arm,Open-label Prospective Trial
Brief Title: Camrelizumab Combined With Apatinib for Advanced Gastric or Esophagogastric Adenocarcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, LiuYing, Deputy Chief Physician, Henan Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-GC-Ⅱ-011
Record Dates: First submitted 2021-06-24; First posted 2021-07-01 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Advanced Gastric Carcinoma
MeSH Terms: interventions — camrelizumab; apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental): camrelizumab combined with apatinib
  Interventions: Drug: camrelizumab; Drug: Apatinib Mesylate

INTERVENTIONS:
Drug: camrelizumab — 200 mg intravenous (IV) camrelizumab on Day 1 and Day 15 of each 28-day cycle.
  Other Names: SHR-1210
Drug: Apatinib Mesylate — 250 mg qd

SUMMARY:
This study is a phase II study, to evaluate the effectiveness and safety of Camrelizumab combined with apatinib for advanced gastric or esophagogastric adenocarcinoma progressed after immune checkpoint inhibitors.

ELIGIBILITY:
Inclusion Criteria:

1. The patient volunteered to participate in the study and signed an informed consent form；
2. ≥18 years old; male or female
3. confirmed incurable gastric and gastroesophageal junction adenocarcinoma（unresectable or metastatic) by pathological examination,at least have a measurable lesion without local treatment.(According to the RECIST V1.1,the long diameter of the lesion can be measured by spiral CT ≥10mm or the short diameter of the enlarged lymph nodes≥15mm;
4. Adequate standard treatment was used in the past; At least two cycles of anti-PD-1 / PD-L1 / CTLA-4 antibody therapy and platinum based chemotherapy were used in the past; Imaging confirmed disease progression occurred during or within 12 weeks after the treatment with anti-PD-1 / PD-L1 / CTLA-4 antibody；
5. It can provide the detection report of human epidermal growth factor receptor 2 (HER2); HER2 negative patients could be included in the study; HER2 positive patients who had failed to receive trastuzumab treatment in the past could be included in the study (HER2 positive was defined as ≥ 10% of tumor cells HER2 IHC 3 + or fish positive)；
6. Swallowing pills normally；
7. ECOG score: 0~1 points;
8. Expected survival period ≥ 12 weeks; A histological specimen can be provided for secondary testing;
9. The main organ function meets the following criteria( It is not allowed to use any blood components or cell growth factor drugs within 14 days before the first medication）:

   The absolute value of neutrophils (ANC) ≥ 1.5 × 109 / L; Platelet (PLT) > 100 × 109 / L ；Albumin(ALB)≥ 90g / L;Total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal (ULN); Alanine aminotransferase (ALT) Aspartate aminotransferase (AST) ≤3 * ULN; serum creatinine (Cr) ≤ 1.5 * ULN ; Thyroid stimulating hormone (TSH) ≤ 1 × ULN (if abnormal, FT3 and FT4 levels should be examined at the same time; if FT3 and FT4 levels are normal, they can be included in the group);Alkaline phosphatase（AKP)≤ 2.5 times the upper limit of normal (ULN).
10. Women of childbearing age should agree to use contraceptives (such as intrauterine devices, contraceptives or condoms) during the study period and within 3 months after the end of the study; negative serum or urine pregnancy test within 72 hours prior to study enrollment and must be non-lactating patients; men should agree to patients who must use contraception during the study period and within 3 months after the end of the study period.

Exclusion Criteria:

1. Any active autoimmune disease or history of autoimmune disease (such as but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hypophysitis, vasculitis, nephritis, hyperthyroidism; Patients with vitiligo or asthma in childhood had complete remission and did not need any intervention in adulthood were included; Asthma requiring medical intervention with bronchodilators could not be included;
2. Those who are using immunosuppressant or systemic hormone therapy to achieve the purpose of immunosuppression (dose > 10mg / day prednisone or other therapeutic hormones) and continue to use them within 2 weeks before entering the group;
3. Severe allergic reaction to other monoclonal antibodies;
4. Patients who end treatment due to related toxicity during anti-PD-1 / PD-L1 / CTLA-4 antibody treatment;
5. Patients with known central nervous system metastasis (except patients with stable disease control and asymptomatic after four weeks of radiotherapy or surgery) or evidence of cancerous meningitis;
6. Squamous or undifferentiated carcinoma of the stomach or gastroesophageal junction;
7. The patients with ascites or pleural effusion with clinical symptoms who need puncture drainage or who have received pleural or ascites drainage within 2 weeks before randomization, except those who only showed a small amount of ascites or pleural effusion without clinical symptoms;
8. Other malignant tumors in the past 3 years or at the same time (except for cured basal cell carcinoma of skin and carcinoma in situ of cervix);
9. Patients with hypertension and cannot be well controlled after antihypertensive drug treatment (systolic pressure ≥ 140 mmHg or diastolic pressure ≥ 90 mmHg);
10. There are clinical symptoms or diseases that can not be well controlled, such as: (1) heart failure of NYHA grade 2 or above (2) unstable angina pectoris (3) myocardial infarction within one year (4) clinically significant supraventricular or ventricular arrhythmias need treatment or intervention (5) QTc > 450ms (male); QTc > 470ms (female);
11. Low dose aspirin and low molecular weight heparin are allowed for prophylactic use in patients undergoing thrombolytic or anticoagulant therapy;
12. In the first 3 months of randomization, there were significant clinical bleeding symptoms or clear bleeding tendency, such as gastrointestinal bleeding, esophageal and gastric varices with bleeding risk, hemorrhagic gastric ulcer or vasculitis; If the fecal occult blood is still positive at baseline (except for weak positive and no clinical significance judged by the researcher), gastroscopy should be performed (the researcher can judge whether gastroscopy should be performed for those who have undergone total gastrectomy before). If the gastroscopy results indicate severe gastric ulcer or the risk of bleeding judged by the researcher, they can not be enrolled; Gastrointestinal perforation or fistula occurred within 3 months before randomization;
13. The events of arteriovenous thrombosis occurred within 6 months before entering the group, such as cerebrovascular accidents (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism, etc;
14. Known hereditary or acquired bleeding and thrombotic tendency (such as hemophilia, coagulation dysfunction, etc.)
15. Urine routine examination showed that urine protein was ≥ +, and 24-hour urine protein> 1.0 g；
16. Those who had received radiotherapy, chemotherapy, surgery (except diagnostic surgery) or trastuzumab for less than 4 weeks before randomization (palliative radiotherapy or local treatment can be extended to 2 weeks before randomization); Or the adverse reactions caused by previous treatment (except hair loss) did not return to ≤ CTCAE 5.0 1level ；
17. Patients with bone metastases received palliative radiotherapy in more than 5% bone marrow area within 2 weeks before the study；
18. Active infection, fever of unknown origin ≥ 38.5 ℃ within 7 days before medication, or white blood cell count > 15 at baseline × 109/L；
19. Congenital or acquired immune deficiency (such as HIV infection)；
20. Active hepatitis (hepatitis B reference: HBsAg positive and HBV DNA > 500 IU/ml); HCV reference: HCV antibody positive and HCV copy number > upper limit of normal value)；
21. Previous treatment with camrelizumab or apatinib;
22. Live vaccine may be vaccinated less than 4 weeks before or during the study;
23. According to the judgment of the researchers, the patients may have other factors that may affect the research results or lead to the termination of the study, such as alcoholism, drug abuse, other serious diseases (including mental illness) requiring combined treatment, serious laboratory abnormalities, family or social factors, which will affect the safety of the patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-04-28 (Actual); Primary Completion 2022-06-03 (Estimated); Study Completion 2023-08-03 (Estimated)

PRIMARY OUTCOMES:
Objective response rate(ORR) | up to 1 years
  ORR was defined as the percentage of participants with best overall response of either CR or PR

SECONDARY OUTCOMES:
Progression-Free Survival(PFS) | up to 2 years
  PFS was defined as the time from the first day of treatment to the first documented disease progression per RECIST 1.1 based on investigator assessment, or death due to any cause, whichever occurs first.
Overall Survival (OS) | up to 2.5 years
  OS was defined as the first day of treatment to death due to any cause.
Disease control rate(DCR) | up to 1 years
  DCR was defined as the percentage of participants with best overall response of either CR or PR or SD
Time to progression(TTP) | up to 2years
  TTP was defined as the time from the first day of treatment to the first documented disease progression per RECIST 1.1 based on investigator assessment in All Participants.
Duration of response(DOR) | up to 2years
  DOR was defined as the time from first documented evidence of CR or PR until disease progression or death due to any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Liu, Principal Investigator — Henan Cancer Hospital
Locations (1):
- Henan cancer hospital/The affiliated Cancer Hospital of ZhengZhou university, Henan, China